CLINICAL TRIAL: NCT01340274
Title: Evaluating the Benefits of the Community Reinforcement and Family Training(CRAFT) Approach to Concerned Significant Others(CSO) of Individuals Engaged in Problem Gambling (IPGs)
Brief Title: Community Reinforcement Approach and Family Training (CRAFT) for Problem Gambling
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Could not get participants
Sponsor: Colchester East Hants Health Authority (Other)
Collaborators: Pictou County Health Authority (Unknown); University of Calgary (Other); Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2011-02-04; First posted 2011-04-22 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2011-04

CONDITIONS: Pathological Gambling
Keywords: Community Reinforcement and Family Training; Concerned Significant Others; Identified Problem Gambler; Therapeutics
MeSH Terms: conditions — Gambling | interventions — Therapeutics; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Usual (Active Comparator): Clients will receive 12 sessions of "Treatment as usual ", delivered 1 session per week for 12 consecutive weeks.
  Interventions: Behavioral: Treatment as Usual
- CRAFT Treatment (Experimental): Clients will receive 12 sessions of "CRAFT", delivered 1 session per week for 12 consecutive weeks.
  Interventions: Behavioral: CRAFT treatment

INTERVENTIONS:
Behavioral: CRAFT treatment — Clients will receive 12 sessions of CRAFT delivered over a 12 week period. There will be 1 session per week.
  Other Names: Community Reinforcement Approach and Family Training
  Arms: CRAFT Treatment
Behavioral: Treatment as Usual — Clients will receive Treatment as Usual delivered over 12 session. There will be 1 session per week.
  Other Names: Cognitive Behavioural Therapy; Motivational Enhancement
  Arms: Treatment as Usual

SUMMARY:
Nova Scotia is experiencing a proliferation of gambling opportunities and their related gambling problems. The 2003 Nova Scotia Prevalence Study (2004) found that approximately 50,000 adult Nova Scotians are at some risk for problem gambling and that approximately 93,000 adult Nova Scotians are intimately connected to at least one person who has a gambling problem. The serious consequences of problem gambling are being felt by the Individuals engaging in Problem Gambling (IPGs), their Concerned Significant Others (CSOs) and their Communities.

Very few IPGs access support services for their gambling problems. Some reports (National Gambling Impact Study Commission 1999) have found that only 3% of IPGs seek treatment. The Nova Scotia Gambling Prevalence Study (2004) states: "Overall, 3.5% (26,000 adults) have been motivated to help someone else with a current gambling problem versus 0.5% (3,700 adults) seeking assistance or information for a personal problem". While the CSOs of IPGs are seven times more likely to access professional addiction treatment the options for these individuals are limited and treatment programs often lack evidence in support of their effectiveness.

The Community Reinforcement and Family Training (CRAFT) (Meyers & Wolfe 2004) approach provides significant benefits to the CSOs of persons abusing alcohol and other drugs. They benefits include: improvement in the quality of life of the CSOs; increasing the rate of substance abusers entering treatment; and decreased substance use. CRAFT empowers CSOs by providing tools to positively influence theirs and their significant other's behavior.

The current study investigates the applicability and effectiveness of the CRAFT approach to the CSOs of IPGS.

It is predicted that benefits to the CSOs receiving CRAFT will significantly surpass those receiving treatment as usual. The predicted benefits are: improvement in quality of life for the CSO; engagement of IPGs in treatment; and decreased gambling by the IPGs. With these achieved outcomes, this research will provide opportunity for earlier intervention, improved individual and family functioning and a reduction of the negative impact of problem gambling on the community.

DETAILED DESCRIPTION:
It has been estimated that 50,000 adult Nova Scotians are at some risk for problem gambling and approximately 93,000 adult Nova Scotians are intimately connected to at least one person who has a gambling problem (Nova Scotia Prevalence Study 2004). The serious consequences of problem gambling are being felt by Individuals engaged in Problem Gambling (IPGs), their Concerned Significant Others (CSOs) and their Communities.

It is known that despite the negative consequence of problem gambling very few IPGs access services for treating their gambling problems. The Nova Scotia Gambling Prevalence Study (2004) has shown that CSOs are seven times more likely to access services than IPGs "Overall, 3.5% (26,000 adults) have been motivated to help someone else with a current gambling problem versus 0.5% (3,700 adults) seeking assistance or information for a personal problem". Despite such findings the treatment options for the CSOs of IPGs are limited (Crisp, B.R. et al. 2001; Shaw, M.C. et al. 2007).

The Community Reinforcement and Family Training (CRAFT) (Meyers & Wolfe 2004) model for CSOs of substance abusers has demonstrated significant success with the following outcomes: improvement in the quality of life of CSOs; engagement of the substance abuser in treatment; and decreased substance use. CRAFT empowers CSOs by providing tools to positively influence their own and their significant others behavior through a cognitive behavioral approach.

This current project investigates the applicability and effectiveness of the CRAFT model as a tool for supporting the CSOs of problem gamblers. A comparative analysis will be completed with random assignment of 60 CSOs to either of Group A (CRAFT) or Group B (treatment as usual). Twelve individual treatment sessions will be offered to each of the CSOs. It is predicted the outcomes of from Group A (CRAFT) will significantly surpass those from Group B (treatment as usual). The predicted outcomes are: improvement in quality of life for the CSOs; engagement of the IPGs in treatment; and decreased gambling by the IPGs. All therapists in the CRAFT experimental group have been certified in the CRAFT model. A comparative analysis will be conducted with the CRAFT approach (Group A) and the traditional treatment approach (Group B). Model adherence will be supervised and tested.

ELIGIBILITY:
Inclusion Criteria:

1. Concerned Significant Other (CSO) must have a significant relationship with the Individuals Engaged in Problem Gambling (IPG)(e.g. parent, child, sibling, friend, partner).
2. CSO must have face-to-face contact with the IPG at least 3 days per week and for at least 1 hour per day with no anticipated relationship change (e.g. separation) over the next 90 days.
3. Impaired functioning of the CSO consequential to their significant other being engaged in problem gambling.
4. Evidence (from the CSOs) that the IPG meets Canadian Problem Gambling Index (CPGI) criteria for problem gambling.
5. The CSO's primary motivation for treatment is to influence their IPG's gambling behaviour.

Exclusion Criteria:

1. CSO meets CPGI criteria for having problem gambling.
2. CSO has a condition, including substance dependency and/or significant psychopathology, which could impede the CSO's ability to understand and participate in treatment.
3. The IPG has received treatment for problem gambling in the previous 3 months, is currently willing to receive treatment, or has been court ordered to receive treatment.
4. Domestic violence is a significant risk based on the CSOs report and psychometric measure.
5. The CSO is currently receiving psychotherapy for issues related to their IPG's gambling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06-03 (Estimated); Primary Completion 2012-04-15 (Actual); Study Completion 2012-04-15 (Actual)

PRIMARY OUTCOMES:
Concerned Significant Other Status (Quality of Life) | Baseline: At 0 weeks
  Measured through the following Tests:
  Beck Depression Inventory (Beck, Steer & Garbin 1988) State/Trait Anxiety Inventory (Speilberger 1999) State-trait Anger Expression Inventory-II (Speilberger et al. 1988) DSM -IV Screening Questionnaire; Social functioning and Resources Scale (Moos et al 1987) Physical symptoms (Moos et al 1987)

SECONDARY OUTCOMES:
Concerned Significant Other Status (Quality of Life) | Post treatment: 1 week
  Measured through the following Tests:
  Beck Depression Inventory (Beck, Steer & Garbin 1988) State/Trait Anxiety Inventory (Speilberger 1999) State-trait Anger Expression Inventory-II (Speilberger et al. 1988) DSM -IV Screening Questionnaire; Social functioning and Resources Scale (Moos et al 1987) Physical symptoms (Moos et al 1987) Significant Other Status (Quality of Life)
Concerned Significant Other Status (Quality of Life) | Follow up: 9 months
  Measured through the following Tests:
  Beck Depression Inventory (Beck, Steer & Garbin 1988) State/Trait Anxiety Inventory (Speilberger 1999) State-trait Anger Expression Inventory-II (Speilberger et al. 1988) DSM -IV Screening Questionnaire; Social functioning and Resources Scale (Moos et al 1987) Physical symptoms (Moos et al 1987)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Purvis, MSc, Principal Investigator — Pictou County Health Authority; David Hodgins, PhD, Principal Investigator — University of Calgary
Locations (3):
- Canada (3):
  - Addiction Services, Amherst, Nova Scotia
  - Addiction Services, Pictou, Nova Scotia
  - Addictions Services, Truro, Nova Scotia